CLINICAL TRIAL: NCT06043271
Title: A Single Session Parenting Intervention Administered to Parents of Children Waiting to Receive Cognitive Behavioral Therapy
Brief Title: A Single Session Parenting Intervention for Children on a Outpatient Therapy Waitlist
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AIM Youth Mental Health (Unknown); American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Madelaine R. Abel, PhD, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001725
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Accommodation; Parenting; Online Intervention; Single Session Intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized (1:1 allocation ratio) to receive the EMPOWER Program single session intervention (SSI) or to have their child remain on the clinic waitlist as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The EMPOWER Program (Experimental): The EMPOWER Program (Sung et al., 2021) is a web-based, self-administered SSI for parents that takes about 30 minutes to complete. The SSI includes 5 elements based on the components of CBT.
  Interventions: Behavioral: The EMPOWER Program
- Waitlist as Usual (No Intervention): Participants in the control group will have their children remain on the waitlist until they are assigned to a therapist in the clinic.

INTERVENTIONS:
Behavioral: The EMPOWER Program — The EMPOWER Program is a web-based, self-administered SSI for parents that takes about 30 minutes to complete.
  Other Names: Project EMPOWER
  Arms: The EMPOWER Program

SUMMARY:
Cognitive Behavioral Therapy (CBT) is the treatment of choice for youth anxiety. However, up to 80% of youth with anxiety disorders do not access the services they need. Child CBT clinics nationwide have extremely long waits, on the order of 10-12 months. This leads to a vicious cycle, as children waiting for care experience worsening symptoms and decreased motivation, so that by the time they access care, their needs are more intensive and the treatment lasts longer and it takes longer for new children to be able to be assigned. Recently, single-session interventions (SSIs) have been developed that enable children to access CBT skills. The proposed randomized trial will evaluate the effects of a brief, web-based, self-guided SSI designed to reduce parent accommodation of children's anxiety, a parenting behavior that has been shown to maintain and worsen child anxiety. The main aim of the study is to examine whether the SSI reduces parent accommodation. As a secondary aim, the investigators will explore whether the SSI reduces children's anxiety symptoms over the first 6 months of CBT. The investigators will recruit parents of children who are on the waitlist to receive outpatient CBT. Results may suggest a promising approach to intervene with parents and children waiting to receive therapy.

DETAILED DESCRIPTION:
Anxiety disorders affect as many as 30% of youth and are associated with academic and social impairment and onset of comorbid mood and substance use disorders. Cognitive Behavioral Therapy (CBT) is the treatment of choice for anxiety, achieving remission rates of 60% alone or 80% in combination with medication. However, up to 80% of youth with anxiety disorders do not access the services they need. CBT clinics nationwide have extremely long waits, on the order of 10-12 months. This leads to a vicious cycle, as children waiting for care experience worsening symptoms and decreased motivation, so that by the time they access care, their needs are more intensive and the treatment lasts longer and it takes longer for new children to be able to be assigned.

One proposed pathway to increase access to mental health services is through the delivery of single session interventions (SSIs). SSIs are defined as structured programs that involve one visit or mental health encounter. SSIs are brief, scalable, and there is extensive evidence demonstrating that they can decrease anxiety among children and adolescents recruited from the general community. Importantly, SSIs can be delivered in a self-guided online format. Thus, they are flexible in delivery and content and uniquely suited to be implemented in an outpatient mental health setting for patients on long outpatient therapy waitlists.

One such SSI is the online, self-guided, EMPOWER Program. This SSI takes 30 minutes and targets parent accommodation, a tendency to facilitate avoidance and enable anxious coping that has been shown to maintain and worsen child anxiety and OCD. This SSI has shown promise in reducing parent accommodation of children's anxiety in non-clinical community samples. However, it has not yet been tested among children seeking psychotherapy services who present with higher acuity. Thus, the goal of this project is to test the EMPOWER SSI delivered to parents of children on the waitlist for outpatient CBT. Parent participants will be randomized to either the SSI or to remain on the waitlist as usual for monitoring. The investigators predict that parents who receive the SSI, compared to the control group, will report (a) greater reductions in accommodation from baseline to 2-week follow-up. As a secondary hypothesis, the investigators will explore whether children of parents who received the SSI will show more rapid improvements in anxiety symptoms over the first 6 months of CBT.

ELIGIBILITY:
Inclusion Criteria:

Parents will be eligible to participate if:

1. Their child has anxiety and/or Obsessive-Compulsive Disorder (OCD) (either subclinical or clinical), as determined by an initial screening
2. Their child is between the age of 5 and 12 years-old
3. Parents are English-speaking
4. Parents are over the age of 18 years old

Exclusion Criteria:

Parents will be excluded if:

1. Their child shows symptoms of suicidal or homicidal ideation, psychosis, or primary severe mood or behavior disorder (i.e., if treatment for another disorder other than anxiety is indicate prior to treatment for anxiety)
2. Their child is already receiving CBT (i.e., transfer cases from other CBT providers in the community).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Accommodation Scale, Parent-Report | Baseline to 2-week follow up
  The Pediatric Accommodation Scale is a parent-report of accommodation of their offspring's anxiety. Parents are asked to rate, on a 5-point scale from 0 (never) to 5 (always), the extent to which they accommodate their child's anxiety or avoidance behaviors. Total scores range from 0 to 25, with higher scores reflecting greater parental accommodation. Parents will report on their accommodation behaviors at baseline and 2-weeks follow-up.

SECONDARY OUTCOMES:
Change in Spence Child Anxiety Scale, Parent-Report Total score | Baseline to 2-week follow up; Change over first 6 months of CBT (intake to 3- and 6-month follow-up)
  The Spence Child Anxiety Scale is a 38 item parent-report assessment of child anxiety symptoms. Parents are asked to rate on a 4-point scale (0-3) the presence of different anxiety symptoms in their children. Items are summed and higher scores reflect more severe child anxiety symptoms. Parents will report on their children's anxiety symptoms at baseline and 2-week follow-up. After children from the waitlist are assigned to a therapist to begin CBT, parents will complete this questionnaire prior to treatment onset (intake), and at 3- and 6-months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No